CLINICAL TRIAL: NCT00645320
Title: An Open Label, Extension Study To Assess The Efficacy And Tolerability Of Oral Ziprasidone In Patients Successfully Completing A Previous Study With Ziprasidone
Brief Title: A Study of Ziprasidone for the Treatment of Psychosis in Patients Who Had Already Had Benefits From Ziprasidone Treatment in a Previous Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281114
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Pyschotic Disorders
MeSH Terms: interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Oral ziprasidone tablets 40 or 80 mg twice daily with meals for 3 months. Doses were flexible based on investigator's discretion.
  Other Names: Geodon, Zeldox

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of ziprasidone in patients who successfully completed a study of ziprasidone treatment of psychosis (Protocol A1281074).

ELIGIBILITY:
Inclusion Criteria:

* Psychotic disorder
* Completion of previous study of intramuscular ziprasidone
* Ability to continue with oral ziprasidone

Exclusion Criteria:

* Concomitant treatment with other anti-psychotic agents within 12 hours prior to the enrollment; for depot agents, a period of two weeks or a cycle, whichever is longer, should occur between the last administration and the patient's enrollment.
* Treatment with antidepressants or mood stabilizers within seven days prior to the enrollment; for MAOIs (monoamine oxidase inhibitors) and moclobemide, this period should be of two weeks; for fluoxetine, five weeks.
* Resistance to conventional psychotic agents. (Resistance is defined as a failure to present a therapeutic response during the acute exacerbation after proper attempts of treatment with marketed antipsychotic agents in two or more occasions during the two years prior to the enrollment in the study.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2003-08; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinical Global Impression-Severity (CGI-S) score | Until Final Visit (within 3 months)

SECONDARY OUTCOMES:
Adverse events | Baseline and Months 1, 2, and 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Brazil (8):
  - Pfizer Investigational Site, RIO de Janeiro RJ, Brazil
  - Pfizer Investigational Site, Fortaleza, Ceará
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Jardim Santa Monica SN, Salvador - BA
  - Pfizer Investigational Site, São Paulo, São Paulo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281114&StudyName=A%20study%20of%20ziprasidone%20for%20the%20treatment%20of%20psychosis%20in%20patients%20who%20had%20already%20had%20benefits%20from%20ziprasidone%20treatment%20in%20a%20previ